CLINICAL TRIAL: NCT05706116
Title: A Controlled Human Infection Study of Orally Administered Trichuris Trichiura Eggs in Naïve Adults
Brief Title: Controlled Human Infection Study of Orally Administered Trichuris Trichiura Eggs in Naïve Adults
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: George Washington University (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CHTI-01-21
Record Dates: First submitted 2022-12-27; First posted 2023-01-31 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-12

CONDITIONS: Whipworm; Trichuriasis; Controlled Human Infection
MeSH Terms: conditions — Trichuriasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Trichuris trichiura Egg Inoculum 150 eggs (Experimental): 150 Trichuris trichiura eggs
  Interventions: Biological: Trichuris trichiura Egg Inoculum
- Trichuris trichiura Egg Inoculum 300 eggs (Experimental): 300 Trichuris trichiura eggs
  Interventions: Biological: Trichuris trichiura Egg Inoculum
- Trichuris trichiura Egg Inoculum 450 eggs (Experimental): 450 Trichuris trichiura eggs
  Interventions: Biological: Trichuris trichiura Egg Inoculum

INTERVENTIONS:
Biological: Trichuris trichiura Egg Inoculum — Trichuris trichiura Egg Inoculum that will be used in this study is manufactured by obtaining T. trichiura eggs from the feces of a chronically infected human volunteer, who is negative for HIV, HBV, and HCV. Fecal material is processed following a qualified standard procedure, and after isolating eggs, they are stored at 2-8oC until use. Controls for the manufacturing process are tests for viability (microscopy of larval hatching), species identification (PCR), and microbial bioburden of the eggs.

SUMMARY:
A Controlled Human Infection Model (CHIM) is being developed to provide early proof-of-concept that experimental infection with the intestinal nematode, Trichuris trichiura, is feasible and safe. The proposed model consists of enrolling consenting, healthy, trichuriasis-naïve adults and challenging them with the investigational product, Trichuris trichiura Egg Inoculum, to assess their ability to result in detectable infection. The proposed study will be a feasibility study that will consist of administering different doses of the Trichuris trichiura Egg Inoculum to healthy adult volunteers to determine the optimal dose (i.e., number of T. trichiura eggs) that is safe, well-tolerated and results in consistent infection.

DETAILED DESCRIPTION:
Open-label, dose-escalation clinical study in healthy, trichuriasis-naïve adults:

Study sites:

* George Washington University, Washington, DC
* Laboratory of Parasitic Diseases, National Institute of Allergy and Infectious Diseases, National Institutes of Health, Bethesda, MD
* Number of participants: up to 18 in 3 cohorts of 6 volunteers each

In Cohort 1, six (6) volunteers will receive an inoculum of 150 embryonated Trichuris trichiura eggs. In Cohort 2, six (6) volunteers will receive an inoculum of 300 embryonated Trichuris trichiura eggs. In the optional Cohort 3, six (6) volunteers will receive an inoculum of 450 embryonated Trichuris trichiura eggs.

The cohorts will be enrolled in a staggered fashion with safety data assessed prior to larval dose escalation. Cohort 2 will be inoculated no earlier than 16 weeks after the last volunteer is inoculated in Cohort 1. The optional Cohort 3 will be inoculated no sooner than 16 weeks after the last volunteer is inoculated in Cohort 2. Cohort 3 will be enrolled only if the tolerability of the experimental infection of Cohort 2 is acceptable and does not result in significant adverse events.

* Egg administration schedule: Study Day 0 (single administration)
* Route: oral
* Doses of T. trichiura Egg Inoculum to be tested: 150, 300 and 450 embryonated eggs (high dose optional)
* Study duration: approximately 10 months per study participant

ELIGIBILITY:
Inclusion Criteria:

1. Males or females between 18 and 45 years, inclusive.
2. Good general health as determined by means of the screening procedures.
3. Available for the duration of the trial (approximately 7.5 months).
4. Willingness to participate in the study as evidenced by signing the informed consent document.

Exclusion Criteria:

1. Pregnancy as determined by a positive urine human choriogonadotropin (hCG) (if female).
2. Participant unwilling to use reliable contraception methods while participating in the study (if female of reproductive potential who is engaging in sexual activity that could lead to pregnancy); being of reproductive potential is defined as not being surgically sterile, abstinent from intercourse with a male partner, in a monogamous relationship with a vasectomized partner, at least 2 years post-menopausal, or determined otherwise by medical evaluation to be sterile.
3. Currently lactating and breast-feeding (if female).
4. Evidence of clinically significant neurologic, cardiac, pulmonary, hepatic, rheumatologic, autoimmune, diabetes, or renal disease by history, physical examination, and/or laboratory studies.
5. Has a diagnosis of schizophrenia, bipolar disease or other major psychiatric condition that would make compliance with study visits/procedures difficult (e.g., subject with psychoses or history of suicide attempt or gesture in the 3 years before study entry, ongoing risk for suicide).
6. Known or suspected immunodeficiency or immunosuppression as a result of an underlying illness or treatment.
7. Laboratory evidence of liver disease (alanine aminotransferase [ALT] greater than 1.25-times the upper reference limit).
8. Laboratory evidence of renal disease (serum creatinine greater than 1.25-times the upper reference limit).
9. Laboratory evidence of hematologic disease (hemoglobin <11.1 g/dl [females] or <12.5 g/dl [males]; absolute leukocyte count <3.4 or >11.0 x 103/mm3; absolute eosinophil count >0.6 x 103/mm3 or platelet count <125 x 103/mm3).
10. Positive fecal occult blood test.
11. Infection with a pathogenic intestinal helminth as determined by stool examination for ova and parasites.
12. History of iron deficiency anemia or laboratory evidence of iron deficiency (serum ferritin concentration below the lower reference limit).
13. Other condition that in the opinion of the investigator would jeopardize the safety or rights of a volunteer participating in the trial or would render the participant unable to comply with the protocol.
14. Volunteer has had medical, occupational, or family problems as a result of alcohol or illicit drug use during the past 24 months.
15. Positive ELISA for hepatitis B surface antigen (HBsAg).
16. Positive confirmatory test for HIV infection.
17. Positive confirmatory test for hepatitis C virus (HCV) infection.
18. Using or intends to continue using oral or parenteral corticosteroids, high-dose inhaled corticosteroids (>800 μg/day of beclomethasone dipropionate or equivalent) or other immunosuppressive or cytotoxic drugs within 30 days of the volunteer's expected enrollment in this study or planned use during the study.
19. Known allergy to albendazole.
20. History of previous infection with T. trichiura or continuous residence for more than 6 months in a T. trichiura-endemic area.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Estimated)
Dates: Start 2025-09-10 (Actual); Primary Completion 2027-10-23 (Estimated); Study Completion 2028-04-30 (Estimated)

PRIMARY OUTCOMES:
Solicited adverse events, graded by severity | Day of CHTI through study Day 182
  Frequency of solicited adverse events, graded by severity, from the day of CHTI through study Day 182.
Serious Adverse Events | Day of CHTI through final study visit on study Day 203
  Frequency of CHTI-related Serious Adverse Events from the time of administration of the T. trichiura Egg Inoculum through the final study visit
Unsolicited adverse events | Day of CHTI through study Day 182
  Frequency of unsolicited adverse events, graded by severity, from the time of CHTI through treatment with albendazole (Day 182)
New-onset chronic medical conditions | Day of CHTI through final study visit on study Day 203
  Frequency of new-onset chronic medical conditions through the final study visit
Adverse Events of Special Interest | Day of CHTI through final study visit on study Day 203
  Frequency of Adverse Events of Special Interest through the final study visit
Adverse events related to abnormal clinical safety laboratory parameter (white blood cell count) values | Day of CHTI through final study visit on study Day 203
  Frequency of clinical safety laboratory adverse events related to abnormal white blood cell count (unit of measure = cells/mm^3)
Adverse events related to abnormal clinical safety laboratory parameter (absolute eosinophil count) values | Day of CHTI through final study visit on study Day 203
  Frequency of clinical safety laboratory adverse events related to abnormal eosinophil count (unit of measure = cells/mm^3)
Adverse events related to abnormal clinical safety laboratory parameter (platelet count) values | Day of CHTI through final study visit on study Day 203
  Frequency of clinical safety laboratory adverse events related to abnormal platelet count (unit of measure = cells/mm^3)
Adverse events related to abnormal clinical safety laboratory parameter (hemoglobin concentration) values | Day of CHTI through final study visit on study Day 203
  Frequency of clinical safety laboratory adverse events related to abnormal hemoglobin concentration (unit of measure = g/dL)
Adverse events related to abnormal clinical safety laboratory parameter (serum creatinine concentration) values | Day of CHTI through final study visit on study Day 203
  Frequency of clinical safety laboratory adverse events related to abnormal serum creatinine concentration (unit of measure = mg/dL)
Adverse events related to abnormal clinical safety laboratory parameter (serum alanine aminotransferase concentration) values | Day of CHTI through final study visit on study Day 203
  Frequency of clinical safety laboratory adverse events related to abnormal serum alanine aminotransferase (ALT) concentration (unit of measure = U/L)

SECONDARY OUTCOMES:
Fecal egg detection | Day of CHTI through study Day 182
  Proportion of participants with detectable T. trichiura eggs, at any time point, in fecal samples, as determined by microscopy using the qualified saline flotation technique
Fecal egg counts | Weeks 12 through 26 post-CHTI
  Fecal egg counts as determined by microscopy using the qualified McMaster method, during Weeks 12 through 26 post-CHTI
T. trichiura DNA in fecal samples | Weeks 12 through 26 post-CHTI
  Levels of T. trichiura DNA in fecal samples, as measured by qPCR, during Weeks 12 through 26 post-CHTI

OTHER OUTCOMES:
Serum cytokine concentrations | Weeks 12 through 26 post-CHTI
  Serum cytokine concentrations during Weeks 12 through 26 post-CHTI
Cytokine concentrations of supernatants after stimulation of peripheral blood mononuclear cells (PBMCs) with T. trichiura antigen | Day of CHTI through final study visit on study Day 203
  Cytokine responses to stimulation with T. trichiura and other microbial antigens for total blood cells and peripheral blood monocytes (PBMCs) from the blood
Fecal microbiome | Day of CHTI through final study visit on study Day 203
  Microbial communities present in the fecal samples by DNA and/or RNA sequencing analyses prior to and after exposure to T. trichiura Egg Inoculum

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - George Washington University Medical Faculty Associates, Washington D.C., District of Columbia
  - NIH Clinical Center, Bethesda, Maryland

IPD SHARING:
Plan to Share IPD: No